CLINICAL TRIAL: NCT07064603
Title: Clinical Evaluation of Tunneled Coronally Advanced Flap (TCAF) Versus Coronally Advanced Flap (CAF) Combined With Connective Tissue Graft in the Treatment of Multiple RT2 Gingival Recession Sites: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of (TCAF) Versus (CAF) Combined With Connective Tissue Graft in the Treatment of Multiple RT2 Gingival Recession Sites
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, may mohamed kamal, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-17-1
Record Dates: First submitted 2025-07-01; First posted 2025-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Gingival Recession, Plastic Surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORONAL ADVANCED FLAP WITH CONNECTIVE TISSUE GRAFT (Active Comparator): The surgical papillae will be elevated using split thickness manner while maintaining the blade in a nearly parallel position to the root.
  * The flap apical to the exposed root will be elevated in a full-thickness The full thickness flap covers the avascular root exposure.
  * The releasing vertical incisions will be elevated protect the underlying bone in the lateral areas of the flap.
  * The part of the flap apical to bone exposure will be elevated by split-thickness, this step will be done so it is possible to move the flap passively in the coronal direction.
  * To permit the coronal advancement of the flap, all muscle insertions present in the thickness of the flap will be eliminated. This will be done by keeping the blade parallel to the external mucosal surface.
  The connective tissue graft, is harvested from the hard palate (donor site) then it will be sutured in the surgical recipient site then covered by the coronal advancement of the flap and suturing it.
  Interventions: Procedure: TCAF
- Tunnel coronal advanced flap with connective tissue graft (Experimental): only one surgical papilla will be elevated. The papilla chosen for incision must be with the least interproximal attachment loss. A slightly divergent vertical incision extending beyond the mucogingival junction then a horizontal incision at a distance equal to the recession depth plus 1 mm apical to the papilla tip. The other papillae integrity is preserved , and will be detached using tunneling miniblades and papilla elevator. The flap will be tunneled till the planned papilla .Connective tissue graft will be harvested the graft will be inserted underneath the flap and tunneled below the non-incised papillae. The TCAF is coronally advanced and stabilized 2 mm above the CEJ with sling and simple interrupted sutures at the level of the papillae and simple interrupted sutures for the vertical incision Further coronal advancement of the tunneled papilla with a suspended suture around the with a composite stop
  Interventions: Procedure: TCAF

INTERVENTIONS:
Procedure: TCAF — tunnel coronal advanced flap

SUMMARY:
the aim of the study is to evaluate the changes in gingival recession depth reduction following, treatment of multiple RT2 recession with tunnel coronal advanced flap in comparison to coronal advanced flap, both combined with connective tissue graft

DETAILED DESCRIPTION:
Several techniques for gingival recession defects have been developed for treatment such as are pedicle soft-tissue graft (rotational flap procedures, advanced flap procedure and tunneling), free soft-tissue graft (epithelialized and subepithelial connective tissue graft) and regenerative procedures (barrier membrane or biologic mediators.

The coronally advanced flap and the tunneling technique are the most commonly performed surgical approaches for treating gingival recessions. Barootchi et al. 2024 conducted a clinical study using tunnel coronal advanced flap technique(TCAF) for treating multiple RT2 gingival recession defects ,in order to combine the advantage of both better access and graft stabilization in CAF and the preservation of the integrity of the papilla and better blood supply to the graft present in tunneling technique. From the previous study it was concluded that the combination of both techniques in the same surgical design can improve both the flap and graft vascularization and enhance clinical, esthetic, and patient-reported outcomes. To our knowledge, there is no conducted randomized clinical trials comparing the tunneled coronally advanced flap technique to the coronally advanced flap for gingival depth reduction in multiple RT2 recessions.

So, this clinical trial aims to address this gap of the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older.
* Multiple adjacent recession defect classified as RT2.
* Patients with healthy systemic condition (Mazzotti et al., 2023).
* An esthetic concern or hypersensitivity associated with GR
* The gingival recessions must have at least 1.5 mm of KTW.
* Presence of an identified CEJ (A step ≤ 1mm of the CEJ level)

Exclusion Criteria:

* Full-mouth plaque and bleeding scores >20 (O'Leary et al., 1972)
* Patients with active periodontal disease;
* Intake of any medications known to affect gingival homeostasis or to interfere with wound healing
* Pregnancy and nursing women
* Smokers: a contraindication for any plastic periodontal surgery (Khuller, 2009).
* Absence of cervical restorations, crowding or malalignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Gingival recession depth reduction (GRD) | ONE YEAR

SECONDARY OUTCOMES:
Percentage of mean root coverage (MRC %) | one year
Percentage of complete root coverage (CRC%) | one year
Gingival Recession width | one year
Keratinized tissue width (KTW) | one year
Probing pocket depth | one year
Root coverage esthetic score | one year
  10 is the ideal esthetic score
  Zero points will be assigned if the final position of the gingival margin is equal or apical to the previous recession depth (failure of root coverage procedure), irrespective of color, the presence of a scar, MTC, or MGJ.
  Zero points will also be assigned when a partial or total loss of interproximal papilla (black triangle) occurred following the treatment
Volumetric soft tissue changes | one year
Post-operative pain | 2 Week post-operative
  Visual Analogue Scale (VAS) with numerical scale from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first 2 weeks postoperatively
Post-operative patient satisfaction | one year
  A 3-item questionnaire will be given to the patients to be answered using a 7-point answer scale for assessing their satisfaction with the whole surgical procedure and the achieved results of the procedure performed.